CLINICAL TRIAL: NCT07268651
Title: The Effect of Proprioceptive Training on Gait Performance and Knee Function in Patients With Anterior Cruciate Ligament Reconstruction
Brief Title: Proprioceptive Training for Gait and Knee Function After Anterior Cruciate Ligament Reconstruction
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Universiti Sains Malaysia (Other)
Responsible Party: Principal Investigator, Shazlin Shaharudin, Associate Professor, Universiti Sains Malaysia
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: USM/JEPeM/KK/25030296
Record Dates: First submitted 2025-11-18; First posted 2025-12-08 (Actual); Last update posted 2025-12-08 (Actual); Status verified 2025-12

CONDITIONS: Anterior Cruciate Ligament Reconstruction
Keywords: Proprioceptive Training; Gait Performance; Knee Function; Joint Position Sense

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control Group (Active Comparator): Participants in this arm will receive a standard rehabilitation program adapted from the Massachusetts General Brigham Sports Medicine Anterior cruciate ligament Reconstruction Rehabilitation Protocol. The rehabilitation sessions will be conducted twice per week. The 12-week program is delivered in four progressive phases focusing on graft protection, restoration of knee range of motion, quadriceps activation, balance, and strengthening exercises. No additional proprioceptive training will be provided in this arm.
  Interventions: Behavioral: Standard Rehabilitation
- Proprioceptive Training Group (Experimental): Participants in this arm will receive a structured 12-week proprioceptive training program in addition to the standard rehabilitation protocol. The proprioceptive training is adapted from validated progressive exercise programs using Swiss balls and BOSU balls, and includes balance, coordination, and neuromuscular control exercises. Training sessions are supervised by a physiotherapist and performed three times per week. The progression follows three stages (initial: weeks 1-5, intermediate: weeks 5-8, advanced: weeks 8-12), with advancement allowed only when exercises can be performed with adequate balance control and without pain.
  Interventions: Behavioral: Standard Rehabilitation; Behavioral: Proprioceptive Training

INTERVENTIONS:
Behavioral: Standard Rehabilitation — A standard rehabilitation program adapted from the Massachusetts General Brigham Sports Medicine Anterior cruciate ligament Reconstruction Rehabilitation Protocol. The program consists of supervised rehabilitation sessions conducted twice per week for 12 weeks. The protocol includes four progressive phases focusing on graft protection, restoration of knee range of motion, quadriceps activation, balance training, and progressive strengthening exercises. No proprioceptive training components are included in this intervention.
Behavioral: Proprioceptive Training — A structured 12-week proprioceptive training program performed in addition to standard rehabilitation. The program is adapted from validated progressive proprioceptive exercise protocols using Swiss balls and BOSU balls. Training sessions are supervised by a physiotherapist and conducted three times per week. Exercises progress through three stages (initial: weeks 1-5, intermediate: weeks 5-8, and advanced: weeks 8-12) and include balance, coordination, and neuromuscular control activities. Participants advance to the next level only when exercises can be performed with adequate balance control and without pain.
  Arms: Proprioceptive Training Group

SUMMARY:
Anterior cruciate ligament reconstruction (ACLR) is commonly performed to restore knee stability after injury, but many patients continue to experience gait abnormalities and reduced knee function during rehabilitation. Proprioceptive training is frequently included in rehabilitation programs to improve joint position sense, neuromuscular control, and movement coordination, yet its specific effects on gait performance and knee function after ACLR are not fully understood.

This study aims to investigate the effects of a 12-week proprioceptive training program on gait performance and knee function in patients who have undergone ACLR. Patients who meet the inclusion criteria will undergo baseline assessments, including gait analysis and knee function tests. They will then participate in a structured 12-week proprioceptive training program as part of their rehabilitation, followed by post-intervention assessments using the same measures.

The primary outcomes include changes in gait performance, such as walking speed, step length, cadence, support time, knee motion, and knee joint angles and moments during walking. Secondary outcomes include changes in knee function, including isokinetic muscle strength, joint position sense, and patient-reported outcomes measured by the Lysholm score and the International Knee Documentation Committee (IKDC) questionnaire. The findings from this study may help to clarify the functional benefits of proprioceptive training and support the development of more targeted and effective rehabilitation strategies for patients recovering from Anterior cruciate ligament (ACL) injuries.

DETAILED DESCRIPTION:
Anterior cruciate ligament reconstruction (ACLR) is widely performed to restore knee stability after injury; however, many patients continue to experience altered gait patterns, reduced neuromuscular control, and functional limitations during rehabilitation. Proprioceptive deficits after Anterior cruciate ligament (ACL) injury and surgery can contribute to impaired movement coordination and knee joint instability, highlighting the importance of proprioceptive training as part of the rehabilitation process.

This study aims to examine the effects of a structured 12-week proprioceptive training program on gait performance and knee function in individuals following ACLR. Participants who meet the eligibility criteria will undergo baseline assessments that include gait analysis, knee range of motion, muscle strength evaluation, joint position sense testing, and patient-reported functional outcomes. After baseline testing, participants will be assigned to one of two groups. The control group will receive a standard rehabilitation program, while the proprioceptive training group will receive the same standard rehabilitation combined with an additional proprioceptive training program.

The standard rehabilitation program is adapted from the Massachusetts General Brigham Sports Medicine ACLR Rehabilitation Protocol, with minor modifications to accommodate available equipment and safety considerations. The 12-week rehabilitation process is divided into four progressive phases (Phase I: 0-2 weeks, Phase II: 3-5 weeks, Phase III: 6-8 weeks, and Phase IV: 9-12 weeks), focusing on graft protection, restoration of knee range of motion, quadriceps activation, and gradual strengthening and functional progression.

The proprioceptive training protocol is adapted from previously validated progressive exercise programs that use unstable surfaces such as Swiss balls and BOSU balls to improve gait performance and knee joint function. Participants in the proprioceptive training group will train three times per week for a total of 12 weeks. The progression of exercises follows three phases (initial: weeks 1-5, intermediate: weeks 5-8, and advanced: weeks 8-12) and includes balance, coordination, and neuromuscular control activities. All sessions are supervised by a physiotherapist, and progression to the next level is allowed only when balance control is stable and exercises can be performed without pain or adverse symptoms.

The primary outcomes of this study focus on gait performance, including measures such as walking speed, step length, cadence, support time, and knee peak flexion and extension angles and moments, as well as knee range of motion during walking. Secondary outcomes include changes in knee function, such as isokinetic muscle strength, joint position sense accuracy, and patient-reported scores using the Lysholm and International Knee Documentation Committee (IKDC) questionnaires.

The results of this study may provide a better understanding of the role of proprioceptive training in improving functional recovery after ACLR. By identifying its effects on gait mechanics and knee function beyond standard rehabilitation alone, this research may support the development of more targeted and effective rehabilitation strategies for individuals recovering from ACL injuries.

ELIGIBILITY:
Inclusion Criteria:

* Adults aged 18-40 years who have undergone primary unilateral anterior cruciate ligament reconstruction (ACLR) using an autograft.
* At least 3 weeks postoperatively and currently engaged in the early-stage rehabilitation phase following ACLR.
* Demonstrate near-full passive knee extension (≤ 5° loss) and at least 90° of passive knee flexion in the operated limb.
* Able to walk independently without assistive devices and perform basic functional tasks (e.g., normal walking, single-leg stance).
* No prior surgery or major injury to the contralateral knee or other lower limb joints.
* No neurological, vestibular, or systemic conditions affecting proprioception, motor control, or physical performance.
* Not currently participating in any structured proprioceptive or neuromuscular training programs.
* Willing and able to comply with the intervention protocol and follow-up, and able to provide written informed consent.

Exclusion Criteria:

* History of revision anterior cruciate ligament surgery, bilateral ACLR, or concurrent reconstruction of other knee ligaments (e.g., posterior cruciate ligament, medial collateral ligament, lateral collateral ligament) in the affected knee.
* Meniscal repair or other intra-articular procedures that restrict knee range of motion beyond 3 weeks postoperatively.
* Diagnosed osteoarthritis, rheumatoid arthritis, or other chronic joint diseases affecting the lower limbs.
* Significant injury, surgery, or persistent pain in the contralateral knee, hip, ankle, or spine that could interfere with training or gait.
* History or current diagnosis of neurological disorders (e.g., stroke, multiple sclerosis, Parkinson's disease) or vestibular dysfunction.
* Any cardiopulmonary or systemic condition that contraindicates structured physical exercise.
* Participation in other structured rehabilitation or proprioceptive training programs within the past 3 weeks.
* Cognitive impairment or psychiatric conditions that may interfere with understanding instructions or complying with the protocol.

Ages: 18 Years to 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 30 (Estimated)
Dates: Start 2025-12 (Estimated); Primary Completion 2026-03 (Estimated); Study Completion 2026-04 (Estimated)

PRIMARY OUTCOMES:
Walking Speed | Baseline and 12 weeks post-intervention
  Walking speed during level walking measured using 3D gait analysis. Unit of measure: meters per second (m/s).
Step Length | Baseline and 12 weeks post-intervention.
  Step length measured during level walking using 3D gait analysis. Unit of measure: meters (m).
Cadence | Baseline and 12 weeks post-intervention.
  Cadence during level walking measured using 3D gait analysis. Unit of measure: steps per minute (steps/min).
Single Support Time | Baseline and 12 weeks post-intervention.
  Single support time of the gait cycle measured using 3D gait analysis. Unit of measure: seconds (s).
Double Support Time | Baseline and 12 weeks post-intervention.
  Double support time of the gait cycle measured using 3D gait analysis. Unit of measure: seconds (s).
Peak Knee Flexion Angle | Baseline and 12 weeks post-intervention.
  Peak knee flexion angle during the stance phase measured using 3D gait analysis. Unit of measure: degrees (°).
Peak Knee Extension Angle | Baseline and 12 weeks post-intervention.
  Peak knee extension angle during the stance phase measured using 3D gait analysis. Unit of measure: degrees (°).
Peak Knee Flexion Moment | Baseline and 12 weeks post-intervention.
  Peak external knee flexion moment measured during walking using 3D gait analysis. Unit of measure: Newton-meters per kilogram (Nm/kg).
Peak Knee Extension Moment | Baseline and 12 weeks post-intervention.
  Peak external knee extension moment measured during walking using 3D gait analysis. Unit of measure: Newton-meters per kilogram (Nm/kg).
Knee Range of Motion | Baseline and 12 weeks post-intervention.
  Total sagittal plane knee range of motion measured during level walking using 3D gait analysis. Unit of measure: degrees (°).

SECONDARY OUTCOMES:
Changes in isokinetic knee muscle strength | Baseline and 12 weeks post-intervention
  Isokinetic muscle strength of the knee flexors and extensors will be measured using an isokinetic dynamometer at angular velocities of 60°/s and 180°/s. Peak torque values for flexion and extension will be recorded. Changes from baseline to week 12 will be analyzed.
Changes in knee joint position sense accuracy | Baseline and 12 weeks post-intervention
  Knee joint position sense will be assessed using a passive joint position reproduction protocol on a Biodex isokinetic dynamometer. Participants will be seated with the hip flexed to approximately 85° and the knee aligned with the dynamometer axis. The device will passively move the lower limb to predetermined target angles (30°, 45°, and 60° of knee flexion) at a constant slow angular velocity (2-5°/s), hold the position for five seconds, and then return the limb to the starting position. With eyes closed and exposed to white noise, participants will indicate when they perceive that the target angle has been reached. The absolute reposition error (degrees) between the target and reproduced angles will be used to represent proprioceptive accuracy, and the variable error (degrees) will be used to quantify intra-trial consistency. Three repetitions will be performed for each target angle, presented in random order.
Change in Lysholm Knee Scoring Scale | Baseline and 12 weeks post-intervention
  Knee function will be evaluated using the Lysholm Knee Scoring Scale. This scale ranges from 0 to 100, with higher scores indicating better knee function. The primary analysis will compare the change in Lysholm score from baseline to 12 weeks post-intervention.
Change in International Knee Documentation Committee Subjective Knee Form Score | Baseline and 12 weeks post-intervention
  Knee function will also be evaluated using the International Knee Documentation Committee Subjective Knee Form. This scale ranges from 0 to 100, with higher scores indicating better subjective knee function. The primary analysis will compare the change in IKDC score from baseline to 12 weeks post-intervention.

CONTACTS AND LOCATIONS:
Overall Officials: Shazlin Shaharudin, PhD, Principal Investigator — Universiti Sains Malaysia
Locations (1):
- Leshan Vocational College, Leshan, Sichuan, China

IPD SHARING:
Plan to Share IPD: No
The individual participant data from this randomized controlled trial on proprioceptive training after anterior cruciate ligament reconstruction will not be shared due to concerns about participant privacy and the lack of an approved institutional framework for public data sharing.